CLINICAL TRIAL: NCT06423014
Title: Smart mHealth Strategy in the Delivery of Behavior Change Techniques for Physical Activity and Health Promotion
Brief Title: Smart mHealth Strategy for Physical Activity and Health Promotion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202303041
Record Dates: First submitted 2024-05-08; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-03

CONDITIONS: Health Behavior Change; Wearable Technology; Chatbot; Social Media; Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Wearable Electronic Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control (No Intervention)
- Wearable devices only (Active Comparator)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with the 1st behavior change technique; Behavioral: Wearable devices with the 2nd behavior change technique; Behavioral: Wearable devices with the 3rd behavior change technique; Behavioral: Wearable devices with the 4th behavior change technique; Behavioral: Wearable devices with the 5th behavior change technique; Behavioral: Wearable devices with all behavior change techniques
- Wearable devices with the 1st behavior change technique (Experimental)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with all behavior change techniques
- Wearable devices with the 2nd behavior change technique (Experimental)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with all behavior change techniques
- Wearable devices with the 3rd behavior change technique (Experimental)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with all behavior change techniques
- Wearable devices with the 4th behavior change technique (Experimental)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with all behavior change techniques
- Wearable devices with the 5th behavior change technique (Experimental)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with all behavior change techniques
- Wearable devices with all behavior change techniques (Experimental)
  Interventions: Behavioral: Wearable devices only; Behavioral: Wearable devices with all behavior change techniques

INTERVENTIONS:
Behavioral: Wearable devices only — self-monitoring
  Arms: Wearable devices only; Wearable devices with all behavior change techniques; Wearable devices with the 1st behavior change technique; Wearable devices with the 2nd behavior change technique; Wearable devices with the 3rd behavior change technique; Wearable devices with the 4th behavior change technique; Wearable devices with the 5th behavior change technique
Behavioral: Wearable devices with the 1st behavior change technique — reminder
  Arms: Wearable devices only
Behavioral: Wearable devices with the 2nd behavior change technique — social support
  Arms: Wearable devices only
Behavioral: Wearable devices with the 3rd behavior change technique — Competition
  Arms: Wearable devices only
Behavioral: Wearable devices with the 4th behavior change technique — Goal-setting
  Arms: Wearable devices only
Behavioral: Wearable devices with the 5th behavior change technique — health coach
  Arms: Wearable devices only
Behavioral: Wearable devices with all behavior change techniques — Self-monitoring, health coach, goal-setting, competition, social support, and reminder
  Arms: Wearable devices only; Wearable devices with all behavior change techniques; Wearable devices with the 1st behavior change technique; Wearable devices with the 2nd behavior change technique; Wearable devices with the 3rd behavior change technique; Wearable devices with the 4th behavior change technique; Wearable devices with the 5th behavior change technique

SUMMARY:
The purpose of this study is to develop a Smart mHealth Strategy that delivers behavior change techniques through wearable physical activity trackers and social media chatbots, including self-monitoring, real-time feedback and reminders, goal-setting, competition and rewards, social support, and health coaching. This study also aims to explore the effect of the Smart mHealth Strategy on the behavioral outcomes and psychological factors of physical activity, and physical and mental health. The study design is a three-stage randomized controlled trial. In each stage, 120 are recruited and randomly assigned to control and experimental groups. Participants are adults with insufficient physical activity and a sedentary lifestyle. The Smart mHealth Strategy uses smartwatches and self-developed chatbots. The constrained dialogue content is designed to finally deliver the six behavior change techniques. Data are collected in the pre-, mid-, and post-tests. The measurement includes self-administered questionnaires, Actigraphy GT9X, Inbody 270S, OMRON HEM-7130, and heart rate variability monitors.

ELIGIBILITY:
Inclusion Criteria:

Adults who is the age of majority, with insufficient physical activity, and a sedentary lifestyle who have smartphones

Exclusion Criteria:

* Individuals' health conditions may affect physical activity in daily living and the experiment, such as disability, serious health problems

  * There are unconventional life plans during the experiment, such as going abroad for vacation, pregnancy, and surgery.

    * Individuals have using experiences in any wearable physical activity trackers in the past six months ④ People who have ever had severe allergies to any wearable device ⑤ Professional athletes or student-athletes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subjective physical activity | up to 12 weeks
  International Physical Activity Questionnaire (IPAQ-SF, MET-minute/week)
Objective physical activity | up to 12 weeks
  Actigraphy GT9X and GT3X (MET-minute/week)
Exercise Benefits/Barriers Scale-Concise (EBBS-C) | up to 12 weeks
  Higher score higher benefits and barriers
Exercise self-efficacy scale (EXSE) | up to 12 weeks
  Higher score higher self-efficacy
Physical Activity Self-Regulation Scale (PASR) | up to 12 weeks
  Higher score higher Self-Regulation
Behavioural Regulation in Exercise Questionnaire (BREQ-3) | up to 12 weeks
  Higher score higher Behavioural Regulation

SECONDARY OUTCOMES:
body composition (Inbody) | up to 12 weeks
  Body mass index (BMI, kg/m^2), skeletal muscle index (SMI, kg/m^2), body fat percentage (%), body fat mass (kg), and fat-free mass (kg)
blood pressure | up to 12 weeks
  Systolic and diastolic blood pressure (mmHg)
heart rate variability | up to 12 weeks
  Total power (TP, 0-0.5 Hz), low-frequency power (LF, 0.04-0.15 Hz), high-frequency power (HF, 0.15-0.40 Hz), the ratio of low frequency to high frequency (LF/HF), and the standard deviation of all normal-to-normal intervals (SDNN)
Depression Anxiety Stress Scale (DASS) | up to 12 weeks
  Higher score worse mental health
World Health Organization Quality of Life Scale (WHOQOL-BREF) | up to 12 weeks
  Higher score higher Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan